CLINICAL TRIAL: NCT04977960
Title: MINECRAFT Study: MINEralcorticoid Receptor Antagonism With CanRenone As eFfective Treatment in Moderate to Severe ARDS in COVID-19, a Phase 2 Clinical Trial.
Brief Title: Efficacy of Canrenone as add-on Treatment in Moderate to Severe ARDS in COVID-19
Acronym: MINECRAFT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Milan (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MINECRAFT
Record Dates: First submitted 2021-07-21; First posted 2021-07-27 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: COVID-19; potassium canrenoate
MeSH Terms: conditions — COVID-19 | interventions — Canrenoic Acid; Canrenone

STUDY DESIGN:
Intervention Model Description: Open label, 1:1 randomized parallel arms, Simon's two stage design, single centre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (No Intervention): Patients randomized to the Reference Group will receive the standard-of-care treatments, according to institutional procedures in force:
  * Dexamethasone i.v. 6 mg die for consecutive 5 days
  * Methylprednisolone i.v. 40 mg bid for consecutive 10 days
  * Low-molecular-weight-heparin i.v. at standardized dose of 70 UI/kg twice
  * Remdesivir i.v. 200 mg in bolus (1st day) then 100 mg die for 4 days; remdesivir will be used only in patients supported with low-flow nasal cannula oxygen or Venturi mask
  * Antibiotic therapy:
    * azithromycin: 500 mg/die per os for 5 days
    * ceftriaxone: 2 g i.v. die for 8 days
- Experimental Group (Experimental): Patients randomized in the Experimental Group will receive canrenone as add-on therapy to standard-of-care treatments. Different starting doses of i.v. canrenone will be administrated in a single or double infusion per day, for 7 days, according to the serum concentration of potassium at randomization
  Interventions: Drug: Potassium Canrenoate

INTERVENTIONS:
Drug: Potassium Canrenoate — potassium canrenoate for 7 days in addition to maximal medical treatment
  Other Names: Canrenone
  Arms: Experimental Group

SUMMARY:
The main aim of the study is to estimate the potential efficacy of i.v. canrenone as add-on therapy on maximal medical treatment versus maximal medical treatment alone in treating moderate-to-severe ARDS due to SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 y.o. Since over eighties are very fragile patients, a lot of confounding unpredictable events may interfere with the trial analyses; thus, these patients will be excluded from this exploratory proof-of-concept trial;
* COVID-19 diagnosis through swab within 14 days from the beginning of symptoms
* Hospitalization for moderate to severe ARDS (as determined by PaO2/FiO2 ≤300 mmHg at admission)
* Serum concentration of potassium ≤4.5 mEq/L
* Consent to participate

Exclusion Criteria:

* Invasive mechanical ventilation
* I.v. hydratation with Darrow's solution or half-strength Darrow's solution underway
* Acute cardiovascular event (acute myocardial infarction, acute ischaemic stroke)
* Current malignant disease
* Creatinine >1.8 mg/dL (for women) and >2.0 mg/dL (for men) or glomerular filtration rate <50 mL/mm
* Systolic blood pressure <110 mmHg and/or diastolic blood pressure <60 mmHg
* Known or suspected hypersensitivity to canrenone
* Hyponatremia
* Anuria
* Familial history of porphyria
* Pregnancy and breastfeeding
* known or suspected hypersensitivity to canrenone
* Inclusion in any other pharmacological clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
in-hospital death | At the event (discharge or death)
  patients discharged to a long-term care facility will be classified as "discharged alive"

SECONDARY OUTCOMES:
Need of invasive mechanical ventilation throughout hospitalization | at discharge or death
  Researchers will record if mechanical ventilation has been required during hospitalization (YES) or not (NO)
Duration of hospitalization for alive patients | From date of randomization until the date discharge or in-hospital death from any cause, whichever came first, assessed up to 48 months
  from randomization to discharge
Drug intolerance | From the date of randomization until three days after the end of IMP administration (10 days after randomization)
  measured as number of AR and SAR
Number of hypotensive events | From the date of randomization until three days after the end of IMP administration (10 days after randomization)
  defined as systolic blood pressure constantly <90 mmHg and diastolic blood pressure constantly <60 mmHg)
Number of hyperkaliemias events | From the date of randomization until three days after the end of IMP administration (10 days after randomization)
  defined as [K+]hematic >5.1 mEq/L
Number of renal failures | From the date of randomization until three days after the end of IMP administration (10 days after randomization)
  defined as eGFR <30 ml/min
Change in Sequential Organ Failure Assessment (SOFA) score from randomization to 7 days after randomization | 7 days after randomization
  A score from 0 (better outcome) to 4 (worst outcome) for six different systems (respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems) will be assessed and recorded in CRF
Change in inflammatory status | at 48 hours and 168 hours (7th day) from randomization
  CRP levels, IL-6, Ddimer and Ferritin
Change in respiratory parameters | at 48 hours and 168 hours (7th day) from randomization
  Heart Rate, Blood Pressure (mmHg), PaO2/FiO2 (mmHg), alveolar-arterial gradient (mmHg)
Changes in features of pulmonary interstitial disease measured by chest X-Ray | at 7 days after randomization
Changes in [K+]hematic, renin, AngII, Ang1-7, Ang1-9, aldosterone and structurally related steroids | at randomization and at 48 and 168 hours (7th day) from randomization
  [K+]hematic will be expressed as mEq/L Plasmatic Renin Activity will be expressed as µUI/mL Hematic Concentration of AngII, Ang1-7, Ang1-9, aldosterone and structurally related steroids will be expressed as ng/mL
Correlation between levels of [K+]hematic, renin, AngII, Ang1-7, Ang1-9, aldosterone and structurally related steroids, at basal level (randomization) and clinical outcomes (in-hospital death, need of invasive mechanical ventilation, SOFA score) | at randomization and at 48 and 168 hours (7th day) from randomization
  [K+]hematic will be expressed as mEq/L Plasmatic Renin Activity will be expressed as µUI/mL Hematic Concentration of AngII, Ang1-7, Ang1-9, aldosterone and structurally related steroids will be expressed as ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vicenzi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico

IPD SHARING:
Plan to Share IPD: No